CLINICAL TRIAL: NCT00064662
Title: Randomized Clinical Trial of the Burch Modified Tanagho and Autologous Fascia Sling Procedures for Women With Predominantly Stress Urinary Incontinence
Brief Title: Comparison of Surgical Procedures to Reduce Urinary Stress Incontinence
Acronym: SISTEr
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: University of Alabama at Birmingham (Other); University of California, San Diego (Other); University of Maryland (Other); University of Pittsburgh (Other); University of Texas (Other); The University of Texas at San Antonio (Other); University of Utah (Other); Beaumont Hospital (Other); Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UITN-RCT (completed)
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Urinary Incontinence
Keywords: Stress urinary incontinence; Surgery
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Burch (Other): The Burch colposuspension
  Interventions: Procedure: Burch Modified Tanagho
- Sling (Other): Pubovaginal sling, using autologous rectus fascia
  Interventions: Procedure: Autologous Fascia Sling

INTERVENTIONS:
Procedure: Burch Modified Tanagho — The Burch colposuspension is a well-established procedure for surgically treating women with stress urinary incontinence. The Burch modified colposuspension suspends the anterior vaginal wall (at the level of the bladder neck) with permanent sutures tied to the iliopectineal ligament.
  Arms: Burch
Procedure: Autologous Fascia Sling — The fascial sling is also a well-established procedure for surgically treating women with stress urinary incontinence. The autologous sling procedure places a harvested strip of rectus fascia transvaginally at the level of the proximal urethra. The fascial strip is secured superiorly to the rectus fascia with permanent sutures
  Arms: Sling

SUMMARY:
The primary aim of this clinical trial is to compare the treatment success for two surgical procedures that are frequently used and have similar cure rates, yet have not been compared directly to each other in a large, rigorously conducted randomized trial. The secondary aims of the trial are to compare other outcomes for the two surgical procedures, including quality of life, sexual function, satisfaction with treatment outcomes, complications, and need for other treatment(s)after surgery. Follow-up will be a minimum of two years and up to four years.

ELIGIBILITY:
* Predominant stress urinary incontinence by self-report,examination and test;
* Urethral hypermobility;
* Eligible for both surgical procedures;
* Ambulatory;
* Not pregnant;
* >12 months post-partum;
* No systemic disease known to affect bladder function;
* No current chemotherapy or radiation therapy;
* No urethral diverticulum, augmentation cytoplasty, or artificial sphincter;
* No recent pelvic surgery;
* Available for follow-up and able to complete study assessments;
* Signed informed consent.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2002-02; Primary Completion 2006-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D. Steers, M.D., Study Chair — University of Virginia
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Beaumont Hospital, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Albo M, Wruck L, Baker J, Brubaker L, Chai T, Dandreo KJ, Diokno A, Goode P, Kraus S, Kusek JW, Lemack G, Lowder J, Steers W; Urinary Incontinence Treatment Network. The relationships among measures of incontinence severity in women undergoing surgery for stress urinary incontinence. J Urol. 2007 May;177(5):1810-4. doi: 10.1016/j.juro.2007.01.032. PMID 17437826
- [Background] Albo ME, Richter HE, Brubaker L, Norton P, Kraus SR, Zimmern PE, Chai TC, Zyczynski H, Diokno AC, Tennstedt S, Nager C, Lloyd LK, FitzGerald M, Lemack GE, Johnson HW, Leng W, Mallett V, Stoddard AM, Menefee S, Varner RE, Kenton K, Moalli P, Sirls L, Dandreo KJ, Kusek JW, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Burch colposuspension versus fascial sling to reduce urinary stress incontinence. N Engl J Med. 2007 May 24;356(21):2143-55. doi: 10.1056/NEJMoa070416. Epub 2007 May 21. PMID 17517855
- [Background] Brubaker L, Chiang S, Zyczynski H, Norton P, Kalinoski DL, Stoddard A, Kusek JW, Steers W; Urinary Incontinence Treatment Network. The impact of stress incontinence surgery on female sexual function. Am J Obstet Gynecol. 2009 May;200(5):562.e1-7. doi: 10.1016/j.ajog.2008.11.017. Epub 2009 Mar 16. PMID 19286143
- [Background] Brubaker L, Stoddard A, Richter H, Zimmern P, Moalli P, Kraus SR, Norton P, Lukacz E, Sirls L, Johnson H; Urinary Incontinence Treatment Network. Mixed incontinence: comparing definitions in women having stress incontinence surgery. Neurourol Urodyn. 2009;28(4):268-73. doi: 10.1002/nau.20698. PMID 19274758
- [Background] Burgio KL, Brubaker L, Richter HE, Wai CY, Litman HJ, France DB, Menefee SA, Sirls LT, Kraus SR, Johnson HW, Tennstedt SL. Patient satisfaction with stress incontinence surgery. Neurourol Urodyn. 2010 Nov;29(8):1403-9. doi: 10.1002/nau.20877. PMID 20976815
- [Background] Chai TC, Albo ME, Richter HE, Norton PA, Dandreo KJ, Kenton K, Lowder JL, Stoddard AM; Urinary Incontinence Treatment Network. Complications in women undergoing Burch colposuspension versus autologous rectus fascial sling for stress urinary incontinence. J Urol. 2009 May;181(5):2192-7. doi: 10.1016/j.juro.2009.01.019. Epub 2009 Mar 17. PMID 19296969
- [Background] FitzGerald MP, Burgio KL, Borello-France DF, Menefee SA, Schaffer J, Kraus S, Mallett VT, Xu Y; Urinary Incontinence Treatment Network. Pelvic-floor strength in women with incontinence as assessed by the brink scale. Phys Ther. 2007 Oct;87(10):1316-24. doi: 10.2522/ptj.20060073. Epub 2007 Aug 7. PMID 17684087
- [Background] Kenton K, Richter H, Litman H, Lukacz E, Leng W, Lemack G, Chai T, Arisco A, Tennstedt S, Steers W; Urinary Incontinence Treatment Network. Risk factors associated with urge incontinence after continence surgery. J Urol. 2009 Dec;182(6):2805-9. doi: 10.1016/j.juro.2009.08.032. Epub 2009 Oct 17. PMID 19837421
- [Background] Kirby AC, Nager CW, Litman HJ, FitzGerald MP, Kraus S, Norton P, Sirls L, Rickey L, Wilson T, Dandreo KJ, Shepherd JP, Zimmern P; Urinary Incontinence Treatment Network. Preoperative voiding detrusor pressures do not predict stress incontinence surgery outcomes. Int Urogynecol J. 2011 Jun;22(6):657-63. doi: 10.1007/s00192-010-1336-5. Epub 2010 Dec 10. PMID 21153471
- [Background] Kraus SR, Markland A, Chai TC, Stoddard A, FitzGerald MP, Leng W, Mallett V, Tennstedt SL; Urinary Incontinence Treatment Network. Race and ethnicity do not contribute to differences in preoperative urinary incontinence severity or symptom bother in women who undergo stress incontinence surgery. Am J Obstet Gynecol. 2007 Jul;197(1):92.e1-6. doi: 10.1016/j.ajog.2007.03.072. PMID 17618773
- [Background] Lemack GE, Krauss S, Litman H, FitzGerald MP, Chai T, Nager C, Sirls L, Zyczynski H, Baker J, Lloyd K, Steers WD; Urinary Incontinence Treatment Network. Normal preoperative urodynamic testing does not predict voiding dysfunction after Burch colposuspension versus pubovaginal sling. J Urol. 2008 Nov;180(5):2076-80. doi: 10.1016/j.juro.2008.07.027. Epub 2008 Sep 18. PMID 18804239
- [Background] Lemack GE, Xu Y, Brubaker L, Nager C, Chai T, Moalli P, Kraus SR, Kerr L, Sirls L, Stoddard A; Urinary Incontinence Treatment Network. Clinical and demographic factors associated with valsalva leak point pressure among women undergoing burch bladder neck suspension or autologous rectus fascial sling procedures. Neurourol Urodyn. 2007;26(3):392-6. doi: 10.1002/nau.20325. PMID 17304525
- [Background] Mallett VT, Brubaker L, Stoddard AM, Borello-France D, Tennstedt S, Hall L, Hammontree L; Urinary Incontinence Treatment Network. The expectations of patients who undergo surgery for stress incontinence. Am J Obstet Gynecol. 2008 Mar;198(3):308.e1-6. doi: 10.1016/j.ajog.2007.09.003. PMID 18313452
- [Background] Markland AD, Kraus SR, Richter HE, Nager CW, Kenton K, Kerr L, Xu Y; Urinary Incontinence Treatment Network. Prevalence and risk factors of fecal incontinence in women undergoing stress incontinence surgery. Am J Obstet Gynecol. 2007 Dec;197(6):662.e1-7. doi: 10.1016/j.ajog.2007.08.062. PMID 18060972
- [Background] Nager CW, Albo ME, Fitzgerald MP, McDermott S, Wruck L, Kraus S, Howden N, Norton P, Sirls L, Varner E, Zimmern P; Urinary Incontinence Treatment Network. Reference urodynamic values for stress incontinent women. Neurourol Urodyn. 2007;26(3):333-40. doi: 10.1002/nau.20348. PMID 17315221
- [Background] Nager CW, Albo ME, Fitzgerald MP, McDermott SM, Kraus S, Richter HE, Zimmern P; Urinary Incontinence Treatment Network. Process for development of multicenter urodynamic studies. Urology. 2007 Jan;69(1):63-7; discussion 67-8. doi: 10.1016/j.urology.2006.08.1118. PMID 17270617
- [Background] Nager CW, FitzGerald M, Kraus SR, Chai TC, Zyczynski H, Sirls L, Lemack GE, Lloyd LK, Litman HJ, Stoddard AM, Baker J, Steers W; Urinary Incontinence Treatment Network. Urodynamic measures do not predict stress continence outcomes after surgery for stress urinary incontinence in selected women. J Urol. 2008 Apr;179(4):1470-4. doi: 10.1016/j.juro.2007.11.077. Epub 2008 Mar 4. PMID 18295276
- [Background] Richter HE, Burgio KL, Brubaker L, Moalli PA, Markland AD, Mallet V, Menefee SA, Johnson HW, Boreham MK, Dandreo KJ, Stoddard AM; Urinary Incontinence Treatment Network. Factors associated with incontinence frequency in a surgical cohort of stress incontinent women. Am J Obstet Gynecol. 2005 Dec;193(6):2088-93. doi: 10.1016/j.ajog.2005.07.068. PMID 16325621
- [Background] Richter HE, Diokno A, Kenton K, Norton P, Albo M, Kraus S, Moalli P, Chai TC, Zimmern P, Litman H, Tennstedt S; Urinary Incontinence Treatment Network. Predictors of treatment failure 24 months after surgery for stress urinary incontinence. J Urol. 2008 Mar;179(3):1024-30. doi: 10.1016/j.juro.2007.10.074. Epub 2008 Jan 18. PMID 18206917
- [Background] Richter HE, Goode PS, Brubaker L, Zyczynski H, Stoddard AM, Dandreo KJ, Norton PA. Two-year outcomes after surgery for stress urinary incontinence in older compared with younger women. Obstet Gynecol. 2008 Sep;112(3):621-9. doi: 10.1097/AOG.0b013e31818187c2. PMID 18757661
- [Background] Sanses TV, Brubaker L, Xu Y, Kraus SR, Lowder JL, Lemack GE, Norton P, Litman HJ, Tennstedt SL, Chai TC. Preoperative hesitating urinary stream is associated with postoperative voiding dysfunction and surgical failure following Burch colposuspension or pubovaginal rectus fascial sling surgery. Int Urogynecol J. 2011 Jun;22(6):713-9. doi: 10.1007/s00192-010-1328-5. Epub 2010 Dec 3. PMID 21128068
- [Background] Steers W, Richter H, Nyberg L, Kusek J, Kraus S, Dandreo K, Chai T, Brubaker L. Challenges of conducting multi-center, multi-disciplinary urinary incontinence clinical trials: experience of the urinary incontinence treatment network. Neurourol Urodyn. 2009;28(3):170-6. doi: 10.1002/nau.20653. PMID 19030190
- [Background] Subak LL, Brubaker L, Chai TC, Creasman JM, Diokno AC, Goode PS, Kraus SR, Kusek JW, Leng WW, Lukacz ES, Norton P, Tennstedt S; Urinary Incontinence Treatment Network. High costs of urinary incontinence among women electing surgery to treat stress incontinence. Obstet Gynecol. 2008 Apr;111(4):899-907. doi: 10.1097/AOG.0b013e31816a1e12. PMID 18378749
- [Background] Tennstedt S; Urinary Incontinence Treatment Network. Design of the Stress Incontinence Surgical Treatment Efficacy Trial (SISTEr). Urology. 2005 Dec;66(6):1213-7. doi: 10.1016/j.urology.2005.06.089. PMID 16360445
- [Background] Tennstedt SL, Fitzgerald MP, Nager CW, Xu Y, Zimmern P, Kraus S, Goode PS, Kusek JW, Borello-France D, Mallett V; Urinary Incontinence Treatment Network. Quality of life in women with stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2007 May;18(5):543-9. doi: 10.1007/s00192-006-0188-5. Epub 2006 Oct 12. PMID 17036169
- [Background] Tennstedt SL, Litman HJ, Zimmern P, Ghetti C, Kusek JW, Nager CW, Mueller ER, Kraus SR, Varner E; Urinary Incontinence Treatment Network. Quality of life after surgery for stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Dec;19(12):1631-8. doi: 10.1007/s00192-008-0700-1. Epub 2008 Aug 6. PMID 18682875
- [Background] Walsh LP, Zimmern PE, Pope N, Shariat SF; Urinary Incontinence Treatment Network. Comparison of the Q-tip test and voiding cystourethrogram to assess urethral hypermobility among women enrolled in a randomized clinical trial of surgery for stress urinary incontinence. J Urol. 2006 Aug;176(2):646-9; discussion 650. doi: 10.1016/j.juro.2006.03.091. PMID 16813912
- [Background] Zimmern P, Nager CW, Albo M, Fitzgerald MP, McDermott S; Urinary Incontinence Treatment Network. Interrater reliability of filling cystometrogram interpretation in a multicenter study. J Urol. 2006 Jun;175(6):2174-7. doi: 10.1016/S0022-5347(06)00343-0. PMID 16697832
- [Background] Zyczynski HM, Lloyd LK, Kenton K, Menefee S, Boreham M, Stoddard AM; Urinary Incontinence Treatment Network (UITN). Correlation of Q-tip values and point Aa in stress-incontinent women. Obstet Gynecol. 2007 Jul;110(1):39-43. doi: 10.1097/01.AOG.0000267190.09976.81. PMID 17601894
- [Background] Kraus SR, Lemack GE, Sirls LT, Chai TC, Brubaker L, Albo M, Leng WW, Lloyd LK, Norton P, Litman HJ; Urinary Incontinence Treatment Network. Urodynamic changes associated with successful stress urinary incontinence surgery: is a little tension a good thing? Urology. 2011 Dec;78(6):1257-62. doi: 10.1016/j.urology.2011.07.1413. Epub 2011 Oct 11. PMID 21996108
- [Background] Kraus SR, Lemack GE, Richter HE, Brubaker L, Chai TC, Albo ME, Sirls LT, Leng WW, Kusek JW, Norton P, Litman HJ; Urinary Incontinence Treatment Network. Changes in urodynamic measures two years after Burch colposuspension or autologous sling surgery. Urology. 2011 Dec;78(6):1263-8. doi: 10.1016/j.urology.2011.07.1411. Epub 2011 Oct 11. PMID 21996105
- [Background] Zimmern PE, Dandreo KJ, Sirls L, Howell A, Hall L, Gruss J, Jesse K, Dickinson T, Prather C. Lessons from a patient experience survey in a randomized surgical trial of treatment of stress urinary incontinence in women. Int Urogynecol J. 2011 Oct;22(10):1273-8. doi: 10.1007/s00192-011-1507-z. Epub 2011 Jul 26. PMID 21789658
- [Background] Kirby AC, Nager CW, Litman HJ, Fitzgerald MP, Kraus S, Norton P, Sirls L, Rickey L, Wilson T, Dandreo KJ, Shepherd J, Zimmern P; Urinary Incontinence Treatment Network. Perineal surface electromyography does not typically demonstrate expected relaxation during normal voiding. Neurourol Urodyn. 2011 Nov;30(8):1591-6. doi: 10.1002/nau.21080. Epub 2011 May 10. PMID 21560157
- [Derived] Brubaker L, Litman HJ, Kim HY, Zimmern P, Dyer K, Kusek JW, Richter HE, Stoddard A; Urinary Incontinence Treatment Network. Missing data frequency and correlates in two randomized surgical trials for urinary incontinence in women. Int Urogynecol J. 2015 Aug;26(8):1155-9. doi: 10.1007/s00192-015-2661-5. Epub 2015 Mar 24. PMID 25800900
- [Derived] Richter HE, Brubaker L, Stoddard AM, Xu Y, Zyczynski HM, Norton P, Sirls LT, Kraus SR, Chai TC, Zimmern P, Gormley EA, Kusek JW, Albo ME; Urinary Incontinence Treatment Network. Patient related factors associated with long-term urinary continence after Burch colposuspension and pubovaginal fascial sling surgeries. J Urol. 2012 Aug;188(2):485-9. doi: 10.1016/j.juro.2012.04.010. Epub 2012 Jun 15. PMID 22704099
- [Derived] Brubaker L, Richter HE, Norton PA, Albo M, Zyczynski HM, Chai TC, Zimmern P, Kraus S, Sirls L, Kusek JW, Stoddard A, Tennstedt S, Gormley EA; Urinary Incontinence Treatment Network. 5-year continence rates, satisfaction and adverse events of burch urethropexy and fascial sling surgery for urinary incontinence. J Urol. 2012 Apr;187(4):1324-30. doi: 10.1016/j.juro.2011.11.087. Epub 2012 Feb 15. PMID 22341290
- [Derived] Brubaker L, Rickey L, Xu Y, Markland A, Lemack G, Ghetti C, Kahn MA, Nagaraju P, Norton P, Chang TD, Stoddard A; Urinary Incontinence Treatment Network. Symptoms of combined prolapse and urinary incontinence in large surgical cohorts. Obstet Gynecol. 2010 Feb;115(2 Pt 1):310-316. doi: 10.1097/AOG.0b013e3181cb86b2. PMID 20093904
- [Derived] Brubaker L, Moalli P, Richter HE, Albo M, Sirls L, Chai T, Kraus SR, Norton P, Chang D, Tennstedt SL. Challenges in designing a pragmatic clinical trial: the mixed incontinence -- medical or surgical approach (MIMOSA) trial experience. Clin Trials. 2009 Aug;6(4):355-64. doi: 10.1177/1740774509339239. Epub 2009 Jul 22. PMID 19625327
- [Derived] Richter HE, Burgio KL, Chai TC, Kraus SR, Xu Y, Nyberg L, Brubaker L. Predictors of outcomes in the treatment of urge urinary incontinence in women. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20(5):489-97. doi: 10.1007/s00192-009-0805-1. Epub 2009 Jan 30. PMID 19183825
- See also: www.uitn.net — http://www.uitn.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2002 and June 2004 at nine study sites, 2,405 women were screened: 556 were ineligible, 1,193 declined or withdrew consent and one died.
Period: Overall Study
Arm/Group | Burch | Sling
Started | 329 | 326
Completed | 255 | 265
Not Completed | 74 | 61
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 57 | 44
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Administratively withdrawn | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Burch | Sling | Total
Number analyzed (Participants) | 329 | 326 | 655
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 289 | 285 | 574
  >=65 years | 40 | 41 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.5) | 51.6 (10.1) | 51.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 326 | 655
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 329 | 326 | 655

OUTCOME MEASURES:

1. Primary Outcome: 24 Month Cumulative Success Rate Computed From Kaplan Meier Time-to-event Analysis (Reported as Percent Success).
Description: Success defined as composite measure including: no self-reported incontinence symptoms reported on the Medical, Epidemiologic, and Social Aspects of Aging Project (MESA) questionnaire, <15g in pad weight during 24 hr pad test, no incontinence episodes on 3-day voiding diary, negative results (no leakage) on provocative stress test at standardized bladder volume, no retreatment for urinary incontinence. Additional treatment for stress urinary incontinence (SUI) includes anti-incontinence surgery, tightening of sling, collagen injections, medication, behavioral treatment, or devices specifically for the treatment of SUI.
Time Frame: Two years
Population: All participants randomized were included in time to event analysis.
Measure: Number (95% Confidence Interval); unit: % success at 24 months
Arm/Group | Burch | Sling
Number analyzed (Participants) | 329 | 326
% success at 24 months | 38 [32 to 44] | 47 [41 to 53]
Statistical Analysis 1: Comparison: Burch vs Sling; Time to event analysis of 24 month success rates. Null hypothesis is that the distributions in the two groups are equal; Test type: Superiority or Other; p = 0.01, Log Rank; Other = 0

2. Primary Outcome: 24 Month Cumulative Stress Specific Success Rates Computed From Kaplan Meier Time-to-event Analysis (Reported as % Success)
Description: Stress-specific success defined by composite measure including: no self-reported symptoms of stress incontinence reported on the Medical, Epidemiologic, and Social Aspects of Aging Project (MESA) questionnaire , negative results (no leakage) on a provocative stress test at standardized bladder volume and no retreatment for stress incontinence Additional treatment for SUI includes anti-incontinence surgery, tightening of sling, collagen injections, medication, behavioral treatment, or devices specifically for the treatment of SUI.
Time Frame: Two years
Population: All participants randomized were included in time to event analysis
Measure: Number (95% Confidence Interval); unit: % stress-specific success at 24 m
Arm/Group | Burch | Sling
Number analyzed (Participants) | 329 | 326
% stress-specific success at 24 m | 49 [43 to 55] | 66 [60 to 71]
Statistical Analysis 1: Comparison: Burch vs Sling; Time to event analysis of cumulative success rates in the two groups. Null hypothesis is that the distributions are equal in the two groups; Test type: Superiority or Other; p < 0.001, Log Rank; Chi-square = 16.2
Statistical Analysis 2: Comparison: Burch vs Sling; Kaplan Meier time-to-event analysis of cumulative success rates. Used Wald test of equality of survival distributions; Test type: Superiority or Other; p < 0.0001, Kalpan Meier (Wald statistic); Other = 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Site principal investigators reported adverse events to the adverse events committee comprised of four investigators who were blinded to site-specific information, including surgeon and study procedure. All adverse events were reviewed by the committee assigned a severity code.
Arm/Group | Burch | Sling
Serious Adverse Events (participants affected / at risk) | 32/329 | 42/326
Other Adverse Events (participants affected / at risk) | 156/329 | 206/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Burch (N=329) | Sling (N=326)
Genitourinary (Renal and urinary disorders) | 18 (22) | 29 (30)
Pelvic pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bleeding (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Wound complication requiring surgical intervention (Injury, poisoning and procedural complications) | 12 (13) | 10 (11)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Respiratory distress requiring intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm requiring reintubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Burch (N=329) | Sling (N=326)
Genitourinary (Renal and urinary disorders) | 105 (203) | 157 (305)
Vascular/ Hematologic (Vascular disorders) | 5 (5) | 9 (9)
Wound complication not requiring surgical intervention (Injury, poisoning and procedural complications) | 62 (69) | 66 (71)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9)
Neurologic (Nervous system disorders) | 6 (6) | 5 (5)
Cardiovascular (Cardiac disorders) | 0 (0) | 2 (2)
Allergic (hives, itching) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Constitutional (General disorders) | 3 (3) | 0 (0)
Dermatologic (rash, erythema) (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 7 (7) | 8 (8)

LIMITATIONS AND CAVEATS:
Patients received care at tertiary care centers which could limit the generalizability of the findings. Patients and providers were aware of treatment assignment which could lead to assessment bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No